CLINICAL TRIAL: NCT06180486
Title: Preoperative Mindfulness Meditation for Total Knee Arthroplasty: A Pilot Study
Brief Title: Mindfulness Meditation Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-2131
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Replacement; Mediation; Feasibility
MeSH Terms: conditions — Negotiating

STUDY DESIGN:
Intervention Model Description: Randomized control trial of two groups, intervention vs waitlist control
Masking Description: Patients, research assistants, surgeons, and anesthesiologists are all unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control: Receive MMI After 90 days (Other): The waitlist control group will allow for comparison of those who had access to the mindfulness meditation intervention (MMI) prior to surgery to those who did not. This group will be given the mindfulness meditation intervention 90 days after their surgery when all study questionnaires are complete. Up until 90-days, they will be asked the same questionnaires as the intervention group aside from the MMI practice survey and the exit survey. They will then be given the exit survey 2 weeks after receiving the MMI. This is done to ensure that both groups receive the potential benefit of the teachings and to deter patient dropout for those interested in the study because of wanting to receive the mindfulness training.
  Interventions: Other: Mindfulness Meditation Intervention
- Intervention: Receive MMI before their day of surgery (Experimental): The intervention group will be given the mindfulness meditation intervention (MMI) 1 week prior to their day of surgery. Up until 90-days, they will be asked the same questionnaires as the waitlist control group, with the addition of the MMI practice survey and the exit survey.
  Interventions: Other: Mindfulness Meditation Intervention

INTERVENTIONS:
Other: Mindfulness Meditation Intervention — The mindfulness intervention is a scripted, ~12min audio recording based on core tenets of mindfulness meditation and contextualized for patients undergoing total knee arthroplasty. It teaches sustained attention on the present, body awareness, acceptance of the body's current state, and transformational strategies to cope with emotional or physical stimuli as they arise. It has been created by the study team based on the teachings of Jon Kabat Zinn (founder of mindfulness meditation) and the PI's history teaching yoga and meditation. Patients will be encouraged to review the audio recording once a week.

SUMMARY:
The goal of this pilot study is to develop a randomized control trial study with sufficient power to definitely address if a preop mindfulness meditation intervention can improve post-total knee arthroplasty mental well-being or physical health compared to controls, and if a preop mindfulness meditation intervention can train resilience. The main questions it aims to answer are:

1. Is this preoperative mindfulness meditation study feasible at Hospital for Special Surgery?
2. Can we estimate a control and intervention group central tendency and variability to be used to determine sample size in future study?
3. Does a preoperative mindfulness meditation interventions improve post-total knee arthroplasty mental well-being or physical health compared to controls? Can preoperative a mindfulness meditation intervention train resilience (as measured by increased resilience score)?

Participants will be randomly assigned to be in the intervention group or the waitlist control group. The intervention group gets the mindfulness mediation intervention prior to their day of surgery, and the control group will be given the mindfulness meditation intervention 90 days after their day of surgery.

The waitlist control group allows for comparison between those who got the mindfulness meditation intervention prior to surgery and those who did not while still offering the potential benefits of the intervention after 90 days.

DETAILED DESCRIPTION:
This study will investigate the effect of a preoperative mindfulness meditation intervention (MMI) on outcomes for total knee arthroplasty (TKA) patients at the Hospital for Special Surgery in a randomized controlled trial. Mindfulness meditation is a practice well-known to psychology research based on sustained attention on the present and a non-judgment of one's current situation. It has been used for numerous psychological issues including stress, anxiety, and depression. This intervention group will be compared against a waitlist control group (patients will be told they are on a waitlist to receive the mindfulness intervention, which will occur after data collection has finished for their group). This control has been utilized in several mindfulness meditation studies.

Measures of anxiety, depression, resilience, pain and pain unpleasantness, and overall physical and mental health will be taken after randomization, but before the intervention (or being told they are on the waitlist). Overall physical and mental health measures will also be taken on the day of surgery and final surveys will be collected at 90 days post-op.

The goal of this pilot study is to develop a randomized control trial study with sufficient power to definitely address if a preop mindfulness meditation intervention can improve post-total knee arthroplasty mental well-being or physical health compared to controls, and if a preop mindfulness meditation intervention can train resilience. The main questions it aims to answer are:

1. Is this preoperative mindfulness meditation study feasible at Hospital for Special Surgery?
2. Can we estimate a control and intervention group central tendency and variability to be used to determine sample size in future study?
3. Does a preoperative mindfulness meditation interventions improve post-total knee arthroplasty mental well-being or physical health compared to controls? Can preoperative a mindfulness meditation intervention train resilience (as measured by increased resilience score)?

Participants will be randomly assigned to be in the intervention group or the waitlist control group. The intervention group gets the mindfulness mediation intervention prior to their day of surgery, and the control group will be given the mindfulness meditation intervention 90 days after their day of surgery.

The waitlist control group allows for comparison between those who got the mindfulness meditation intervention prior to surgery and those who did not while still offering the potential benefits of the intervention after 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing primary total knee arthroplasty with a participating surgeon
* Patients on these medications for anxiety/depression: Fluoxetine, Paroxetine, Citalopram, Escitalopram, Sertraline, Fluvoxamine, Venlafaxine, Duloxetine, Levomilnacipran, Desvenlafaxine, Bupropion, Mirtazapine, Amitriptyline, Nortriptyline, Clonazepam, Alprazolam, Lorazepam, Diazepam, Oxazepam, Chlordiazepoxide
* Patients receiving intraoperative auricular acupuncture as part of participating surgeon's preferred anesthetic care
* Patients fluent in English
* ASA I-III
* BMI < 40

Exclusion Criteria:

* Patient not fluent in English (inability to understand the intervention video will likely affect ability to utilize the mindfulness techniques taught)
* Pediatric patients < 18 years of age
* Patients with contraindications to intra-op protocol
* Patients with contraindications to auricular acupuncture (non-native ear, active ear infection, gauges in the ears)
* Patients unable/unwilling to participate in the questionnaires or view the scripted intervention
* Patients scheduled for consecutive or staged surgeries
* Patients allergic to local anesthetics or study medications
* Patients who have kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Overall mental health score | 1 week prior to surgery to post operative day 90
  PROMIS Mental Health Questionnaire is to assess general mental health in patients 1 week prior to surgery, post operative day 14, and post operative day 90. The responses to these questionsare excellent, very good, good, fair, or poor.
Anxiety | 1 week prior to surgery to post operative day 90
  Generalized Anxiety Disorder Assessment (GAD-7) is used to assess severe anxiety in patients 1 Week prior to surgery, post operative day 14, and post operative day 90. The responses to these questions are not at all sure, several days, over half the days, or nearly every day.
Depression | 1 week prior to surgery to post operative day 90
  The Patient Health Questionnaire (PHQ-9) is to assess depression in patients 1 week prior to surgery, post operative day 14, and post operative day 90. The responses to these questions are not at all, Several days, more than half the days, and nearly every day.
Overall physical health scores | 1 week prior to surgery to post operative day 90
  PROMIS Physical Health Questionnaire is used to assess general physical health in patients 1 week prior to surgery, post operative day 14, and post operative day 90. The responses to these questions are excellent, very good, good, fair, or poor.
Knee health | 1 week prior to surgery to pre operative holding
  The KOOS-JR questionnaire will assess knee health after a total knee replacement surgery 1 week prior to surgery, post operative day 14, and post operative day 90. The responses to these questions are none, mild, moderate, severe, or extreme.
MMI Practice Survey | pre-operative holding to post-operative day 90
  The mindfulness meditation intervention practice survey helps to assess enrollment, retention, intervention completion and use measured by time to full enrollment, dropout number/proportion, number of MMI views/uses. The MMI practice survey is asked to the intervention group in pre-operative holding, post-operative day 14 and post-operative day 90. There are several different responses to these questions. These responses include yes or no; from 1-5+; emotional destress or physical pain; Not at all, somewhat improved, improved, or greatly improved.
Exit Survey | pre-operative holding to post-operative day 90
  The exit survey is used to assess ease and helpfulness of the mindfulness meditation intervention to the patients. This is asked to the intervention group in pre-operative holding, post-operative day 14 and post-operative day 90. This survey includes several different respnses to its questions. Responses include; open ended responses; yes or no; < 1 week, 1-2 weeks, 3-4 weeks, or 4+ weeks.

SECONDARY OUTCOMES:
Pain outcomes of patients | 1 week prior to surgery to post operative day 90
  The Pain Unpleasantness scale uses verbal descriptors to asses pain at 1 week prior to surgery, day of surgery, post-acute care unit (PACU), post operative day 14, and post operative day 90. The response to this questionnaire are slightly unpleasant, slightly annoying, unpleasant, annoying, slightly, distressing, very unpleasant, distressing, very annoying, slightly intolerable, very distressing, intolerable, or very intolerable.
Numerical Rating Scale (NRS) | 1 week prior to surgery to post operative day 90
  The NRS assesses pain levels on a scale from 0-10 in the operative knee 1 week prior to surgery, day of surgery, post-acute care unit (PACU), post operative day 14, and post operative day 90.
Resilience training | 1 week prior to surgery to post operative day 90
  The Brief Resilience Scale is used to assess the ability to recover from stress 1 Week prior to surgery, post operative day 14, and post operative day 90. The responses to this questionnaire are strongly agree, disagree, neutral, agree, strongly agree.
Patient satisfaction | Post operative day 14
  The patient satisfaction survey will assess patient satisfaction with results of the total knee replacement surgery taken on post operative day 14. The responses to this questionnaire range from 0-10, 0 being strongly dissatisfied and 10 being strongly satisfied.
Pain catastrophizing scale | 1 week prior to surgery
  The pain catastrophizing scale assess pain experience and ability to cope with pain 1 week prior to surgery. The responses to this questionnaire are not at all, to a slight degree, to a moderate degree, to a great degree, or all the time.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Li, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng SI, Kelleher DC, DeMeo D, Zhong H, Birch G, Ast MP. Intraoperative Acupuncture as Part of a Multimodal Analgesic Regimen to Reduce Opioid Usage After Total Knee Arthroplasty: A Prospective Cohort Trial. Med Acupunct. 2022 Feb 1;34(1):49-57. doi: 10.1089/acu.2021.0072. Epub 2022 Feb 14. PMID 35251437
- [Background] Denkova E, Zanesco AP, Rogers SL, Jha AP. Is resilience trainable? An initial study comparing mindfulness and relaxation training in firefighters. Psychiatry Res. 2020 Mar;285:112794. doi: 10.1016/j.psychres.2020.112794. Epub 2020 Jan 16. PMID 32078885
- [Background] Hanley AW, Gililland J, Erickson J, Pelt C, Peters C, Rojas J, Garland EL. Brief preoperative mind-body therapies for total joint arthroplasty patients: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1749-1757. doi: 10.1097/j.pain.0000000000002195. PMID 33449510
- [Background] Hirschmann MT, Testa E, Amsler F, Friederich NF. The unhappy total knee arthroplasty (TKA) patient: higher WOMAC and lower KSS in depressed patients prior and after TKA. Knee Surg Sports Traumatol Arthrosc. 2013 Oct;21(10):2405-11. doi: 10.1007/s00167-013-2409-z. Epub 2013 Jan 29. PMID 23358576
- [Background] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Background] Jones AR, Al-Naseer S, Bodger O, James ETR, Davies AP. Does pre-operative anxiety and/or depression affect patient outcome after primary knee replacement arthroplasty? Knee. 2018 Dec;25(6):1238-1246. doi: 10.1016/j.knee.2018.07.011. Epub 2018 Aug 16. PMID 30121151
- [Background] Judge A, Arden NK, Cooper C, Kassim Javaid M, Carr AJ, Field RE, Dieppe PA. Predictors of outcomes of total knee replacement surgery. Rheumatology (Oxford). 2012 Oct;51(10):1804-13. doi: 10.1093/rheumatology/kes075. Epub 2012 Apr 24. PMID 22532699
- [Background] Kwak S, Lee TY, Jung WH, Hur JW, Bae D, Hwang WJ, Cho KIK, Lim KO, Kim SY, Park HY, Kwon JS. The Immediate and Sustained Positive Effects of Meditation on Resilience Are Mediated by Changes in the Resting Brain. Front Hum Neurosci. 2019 Mar 26;13:101. doi: 10.3389/fnhum.2019.00101. eCollection 2019. PMID 30983980
- [Background] Magaldi RJ, Staff I, Stovall AE, Stohler SA, Lewis CG. Impact of Resilience on Outcomes of Total Knee Arthroplasty. J Arthroplasty. 2019 Nov;34(11):2620-2623.e1. doi: 10.1016/j.arth.2019.06.008. Epub 2019 Jun 12. PMID 31278038
- [Background] Sharma AK, Elbuluk AM, Gkiatas I, Kim JM, Sculco PK, Vigdorchik JM. Mental Health in Patients Undergoing Orthopaedic Surgery: Diagnosis, Management, and Outcomes. JBJS Rev. 2021 Jul 23;9(7). doi: 10.2106/JBJS.RVW.20.00169. PMID 34297704
- [Background] Singh JA, Yu S, Chen L, Cleveland JD. Rates of Total Joint Replacement in the United States: Future Projections to 2020-2040 Using the National Inpatient Sample. J Rheumatol. 2019 Sep;46(9):1134-1140. doi: 10.3899/jrheum.170990. Epub 2019 Apr 15. PMID 30988126
- [Background] Vissers MM, Bussmann JB, Verhaar JA, Busschbach JJ, Bierma-Zeinstra SM, Reijman M. Psychological factors affecting the outcome of total hip and knee arthroplasty: a systematic review. Semin Arthritis Rheum. 2012 Feb;41(4):576-88. doi: 10.1016/j.semarthrit.2011.07.003. Epub 2011 Oct 28. PMID 22035624
- [Background] Wylde V, Trela-Larsen L, Whitehouse MR, Blom AW. Preoperative psychosocial risk factors for poor outcomes at 1 and 5 years after total knee replacement. Acta Orthop. 2017 Oct;88(5):530-536. doi: 10.1080/17453674.2017.1334180. Epub 2017 May 31. PMID 28562150

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT06180486/Prot_SAP_000.pdf